CLINICAL TRIAL: NCT04498780
Title: Hemodynamic Effects of Angiotensin Receptor Neprilysin Inhibition on Noninvasive Pressure-volume Analysis in Patients With Heart Failure With Reduced Ejection Fraction
Brief Title: Hemodynamic Effects of ARNI on Noninvasive Pressure-volume Analysis in Patients With Chronic Heart Failure
Acronym: ARNI-PVA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Daniel Lavall, Dr. med. Daniel Lavall, University of Leipzig
Other Study IDs: DL-L-20005_V1.4
Record Dates: First submitted 2020-07-29; First posted 2020-08-04 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Heart Failure With Reduced Ejection Fraction
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Sacubitril-Valsartan — Observational study during the clinically indicated treatment

SUMMARY:
Sacubitril-Valsartan reduced heart failure hospitalizations and cardiovascular mortality compared to enelapril in chronic heart failure. Furthermore, quality of life is improved. The decrease of NT-proBNP levels during Sacubitril-Valsartan treatment is associated with reverse left ventricular remodeling and improved left ventricular systolic function. However, the underlying mechanisms that contribute to these symptomatic and prognostic benefits are largely unknown. The aim of this study is to evaluate left ventricular hemodynamics in patients treated with Sacubitril-Valsartan using non-invasive pressure-volume analysis.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic heart failure (NYHA functional class II to IV)
* Reduced LV ejection fraction (≤ 40%)
* Clinical indication for therapy with Sacubitril-Valsartan

Exclusion Criteria:

* catecholamine therapy at inclusion
* existing therapy with Sacubitril-Valsartan
* planned cardiac resynchronization therapy (CRT) within 6 months; inclusion at least 3 months after CRT
* planned mitral or aortic valve procedure within 6 months; inclusion at least 3 months after valve procedure
* participation in another randomized heart failure trial
* severe aortic or mitral valve lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic heart failure (NYHA functional class II to IV) and reduced ejection fraction (LVEF≤40%) with clinical indication for therapy with Sacubitril-Valsartan
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular contractility, afterload and ventricular-arterial coupling | 6 months
  Change of end-systolic elastance (Ees), arterial elastance (Ea) and ventricular-arterial coupling (Ea/Ees)

SECONDARY OUTCOMES:
Systolic and diastolic LV function, symptom status and biomarkers | 3, 6 and 12 months
  * Echocardiography: Left ventricular (LV) remodeling und function (LVEDV, LVESV, LVEF, GLS), diastolic LV function (LAESV, E/e', LVEDP)
  * Symptoms: NYHA functional class, 6 minute walk test
  * Biomarker: NT-proBNP
Left ventricular contractility, afterload and ventricular-arterial coupling | 3 and 12 months
  Change of end-systolic elastance (Ees), arterial elastance (Ea) and ventricular-arterial coupling (Ea/Ees)

OTHER OUTCOMES:
Load-independent parameters of systolic and diastolic LV function, myocardial work indices | 3, 6 and 12 months
  * Peak power index (PPI)
  * Preload-recruitable stroke work (PRSW)
  * End-systolic meridional wall stress (EsMWS)
  * Total peripheral resistance (TPR)
  * LV end-systolic pressure (LVEDP)
  * LV end-diastolic pressure-volume relationship (LVEDPVR)
  * Pressure-strain loops

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lavall, MD, Principal Investigator — University of Leipzig
Locations (2):
- Germany (2):
  - University of Leipzig, Leipzig, Saxony
  - Kardiopraxis Schirmer, Kaiserslautern